CLINICAL TRIAL: NCT01472328
Title: Effects of HBO Therapy on Muscular Insulin Resistence in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Diabetes Center (Other)
Collaborators: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: ROS Paradoxon
Record Dates: First submitted 2011-11-13; First posted 2011-11-16 (Estimated); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Obesity; Non-insulin-dependent Diabetes Mellitus
Keywords: Oxidative stress; Insulin resistance
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Oxidative Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyperbaric oxygen therapy (Experimental): Effect of 2 hrs HBO therapy on muscular insulin sensitivity and resistance in obesity and type 2 diabetes mellitus
  Interventions: Procedure: HBO therapy
- Hyperbaric room air (Sham Comparator): Effect of 2 hrs hyperbaric room air herapy on muscular insulin sensitivity and resistance in obesity and type 2 diabetes mellitus
  Interventions: Procedure: Hyperbaric room air

INTERVENTIONS:
Procedure: HBO therapy — Effect of 2 hrs HBO therapy on muscular insulin sensitivity and resistance in obesity and type 2 diabetes mellitus
  Other Names: oxidative stress; antioxidative capacity
  Arms: Hyperbaric oxygen therapy
Procedure: Hyperbaric room air — Effect of 2 hrs hyperbaric room air on muscular insulin sensitivity and resistance in obesity and type 2 diabetes mellitus
  Other Names: HBO therapy; oxidative stress
  Arms: Hyperbaric room air

SUMMARY:
Hyperbaric oxygen therapy (HBO) is applied for several diseases. The effect on insulin sensitivity is yet unknown. Hypothesis: HBO therapy improves insulin sensitivity in patients.

DETAILED DESCRIPTION:
HBO therapy is applied to improve wound healing in diabetic patients with foot ulcera. However, it might induce oxidative stress as well as improve antioxidative capacity. The effects on insulin sensitivity in humans and will be tested in the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 30 years- ≤ 70 years
* Balanced sex (50: 50)
* BMI 20- 25 kg/m 2 normal- weight group
* BMI 35- 39,9 kg/m 2 (Obese typ II)

Exclusion Criteria:

* Acute illness 2 weeks before start of examination
* Autoimmune or Immune disorder deseases (Leukozyten < 5000/µl
* Renal insufficiency (Kreatin > 1,5 mg/dl)
* Heart disease, condition after heart attack
* Anemia (Hb <12g/l, contolled before every day of eximination) or blood donations 4weeks before eximinatin.
* Participation in another trial within the last 2 weeks
* Pharmacological- immuno therapy (Cortisol, Antihistaminika, ASS)
* Thyroid disorders
* Glitazone or Insulin- Therapy
* Pragnancy, Lactation, Menstruation
* Smoking cigaretts, Alcohol- and drug abuse
* Psychiatric disorders
* Risk for/ or diagnosed HIV/ AIDS or Hepatitis B/C
* Liver disease, which are not caused by non- alcoholic steato- hepatitis
* Working on night shifts or irregular rhythem of night- day
* Impaired wound healing or clotting disorders
* Allergic reaction to local anesthetics
* Malignant cancer

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle insulin sensitivity | 2 years
  Determination of the influence of 2 hours hyperoxygenation on insulin sensitivity redox balance and lipid metabolites of skeletal muscle in patients with T2DM

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, Prof., MD, Principal Investigator — German Diabetes Center
Locations (1):
- German Diabetes Center, Düsseldorf, Germany

REFERENCES:
- See also: Homepage — https://ddz.de/